CLINICAL TRIAL: NCT05858931
Title: Association Between Hysteroscopic Evaluation and the Clinical Outcomes of Vaginal Repair of Cesarean Section Scar Defects
Brief Title: Hysteroscopic Evaluation and the Clinical Outcomes of Vaginal Repair of Cesarean Section Scar Defects
Acronym: CSD
Status: Not yet recruiting | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-23-008
Record Dates: First submitted 2023-05-05; First posted 2023-05-15 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2023-05

CONDITIONS: Magnetic Resonance Imaging; Hysteroscopy
Keywords: cesarean section scar defect; hysteroscopy; surgical outcomes

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CSD patients: All women suffered from abnormal uterine bleeding and were evaluated in a standardized way with hysteroscopy before vaginal surgery.
  Interventions: Procedure: vaginal repair

INTERVENTIONS:
Procedure: vaginal repair — vaginal repair

SUMMARY:
Cesarean section scar defects (CSDs) are one of the long-term complications following cesarean section. They can be detected by transvaginal sonography, hysterosalpingography, sonohysterography and magnetic resonance imaging (MRI). Hysteroscopy is frequently used in evaluating endometrial disease. However, the description of CSDs by hysteroscopy is very limited. Only a few papers about hysteroscopy evaluation have been published. This is an exploratory study to compare hysteroscopic findings with the clinical outcomes of vaginal repair of CSDs.

DETAILED DESCRIPTION:
All women with CSD suffered from abnormal uterine bleeding and were evaluated in a standardized way with hysteroscopy before vaginal surgery. Dome-shaped CSDs could be clearly observed in all patients under hysteroscopy. We recorded the pictures of each patient under hysteroscopy and classified them. They all underwent vaginal excision and suture of CSD and will be required to undergo examinations at 3- and 6-months after surgery. Preoperative and postoperative clinical information will be collected. All patients obtain menstrual information and CSD scar size by MRI or transvaginal sonography.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are non-pregnant patients who had one or more cesarean sections, patients who had intermenstrual spotting after the cesarean section or those in which the TRM was less than 3.0 mm at the preoperative stage, and patients who underwent MRI and TVS to evaluate the size of the defect and the TRM before surgery

Exclusion Criteria:

* Patients who had a history of chronic diseases (such as cerebro-cardiovascular diseases, malignancies and diabetes mellitus), endocrine disorders, menstrual irregularities before cesarean section, coagulation disorders, use of intrauterine devices, sub-mucous myoma, endometrial diseases, endometrial cysts, uterine fibroids, and adenomyosis after cesarean section

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Non-pregnant patients who had one or more cesarean sections, patients who had intermenstrual spotting after the cesarean section or those in which the TRM was less than 3.0 mm at the preoperative stage
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
the days of duration of menstruation | on Days: 1 month
  duration of menstruation
the days of duration of menstruation | on Days: 3 month
  duration of menstruation
the days of duration of menstruation | on Days: 6 month
  duration of menstruation
The thickness of the residual myometrium | on Days: 3-6 month
  The thickness of the residual myometrium

SECONDARY OUTCOMES:
number of pregnancy | 3 years
  reproductive information by questionnaire, including abortion, delivery, childbirth, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Xipeng Wang, Docter, Principal Investigator — Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine

IPD SHARING:
Plan to Share IPD: No